CLINICAL TRIAL: NCT01174407
Title: Is CD35, CD21 and CD55 Associated With Exudative Age-related Macular Degeneration
Brief Title: Implication of CD35, CD21 and CD55 in Exudative Age-related Macular Degeneration
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rudolf Foundation Clinic (Other)
Responsible Party: Prof. Dr. Susanne Binder, Rudolf Foundation Clinic
Other Study IDs: EK08010-VK
Record Dates: First submitted 2008-11-19; First posted 2010-08-03 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-08

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Receptors, Complement 3d; CD55 Antigens

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cd35
  Interventions: Other: cd 35, cd21, cd55

INTERVENTIONS:
Other: cd 35, cd21, cd55 — Blood drawing/ 10ml/ once- duration of 1 day of full examination of the patient

SUMMARY:
The purpose of this study is to determine a possible implication of CD21, CD35 and CD55 in the pathogenesis of age-related macular degeneration. The aim is to asses a difference in expression rates of these factors on AMD-patients and a healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* Man and women over 18 years old
* Filled out informed consent
* Diagnosis of non-exudative/ exudative age related macular degeneneration

Exclusion Criteria:

* Inherited retinal diseases
* Other acquired retinal/ macular
* Missing informed consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with exudative age-related macular degeneration, over 55
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-12 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
determine a possible implication of CD21, CD35 and CD55 in the pathogenesis of age-related macular degeneration | 1 day

SECONDARY OUTCOMES:
expression rates of on AMD-patients and a healthy control group | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Rudolf Foundation Clinic, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Haas P, Aggermann T, Nagl M, Steindl-Kuscher K, Krugluger W, Binder S. Implication of CD21, CD35, and CD55 in the pathogenesis of age-related macular degeneration. Am J Ophthalmol. 2011 Sep;152(3):396-399.e1. doi: 10.1016/j.ajo.2011.02.017. Epub 2011 Jun 12. PMID 21669404